CLINICAL TRIAL: NCT03226080
Title: Combined General and Spinal Anesthesia vs. Combined General and Spinal Anesthesia With Neuromuscular Blockade for Operative Repair of Hip Fractures
Brief Title: GA/Spinal vs. GA/Spinal/NMB for Operative Repair of Hip Fracture
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated with IRB on 20Feb2019 due to lack of enrollment.
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Scott Byram MD, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 209397
Record Dates: First submitted 2017-05-01; First posted 2017-07-21 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Hip Fractures; Anesthesia, Spinal; Anesthesia, General; Neuromuscular Blockade
MeSH Terms: conditions — Hip Fractures | interventions — Rocuronium; Sugammadex; Saline Solution

STUDY DESIGN:
Intervention Model Description: 84 patient under GA with spinal anesthesia will be block randomized to either neuromuscular blockade or placebo. Randomization will be tracked by the research pharmacist at Loyola University
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators, surgeons, intraoperative anesthesiology providers, and patients will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will be monitored and then sedated with midazolam, fentanyl, and ketamine as necessary per standard practice to facilitate lateral positioning. Patients will be positioned with the operative side down for the spinal blockade. Under sterile conditions, spinal anesthesia will be induced with 9mg (1.2mL) of hyperbaric 0.75% bupivacaine as per standard practice. The patient will then be given a standard general anesthetic induction consisting of propofol, succinylcholine, fentanyl, and lidocaine. At the time of incision, this group will be given 10cc normal saline. Once skin closure has been initiated, 2mL normal saline will be administered.
  Interventions: Drug: Normal saline
- Neuromuscular Blockade (Active Comparator): Patients will be monitored and then sedated with midazolam, fentanyl, and ketamine as necessary per standard practice to facilitate lateral positioning. Patients will be positioned with the operative side down for the spinal blockade. Under sterile conditions, spinal anesthesia will be induced with 9mg (1.2mL) of hyperbaric 0.75% bupivacaine as per standard practice. The patient will then be given a standard general anesthetic induction consisting of propofol, succinylcholine, fentanyl, and lidocaine. At the time of incision, this group will be given IV rocuronium 0.6mg/kg in a volume of 10cc. Once skin closure has been initiated, sugammadex 200mg in 2ml will be administered.
  Interventions: Drug: Rocuronium; Drug: Sugammadex

INTERVENTIONS:
Drug: Rocuronium — The neuromuscular blockade group will receive intravenous rocuronium
  Arms: Neuromuscular Blockade
Drug: Sugammadex — The neuromuscular blockade group will receive intravenous sugammadex for reversal of residual rocuronium
  Arms: Neuromuscular Blockade
Drug: Normal saline — Normal saline will be administered as a placebo in equal volume for the placebo group
  Arms: Placebo

SUMMARY:
Surgical repair of hip fractures may be performed with various anesthetic techniques, but are most commonly completed under general anesthesia (GA) or neuraxial anesthesia (NA). Numerous prospective and retrospective studies demonstrate improved morbidity and mortality when NA is used; however, many surgeons prefer the use of GA with neuromuscular blockade (NMB) due to the perception of better operative conditions. This study aims to compare the operative conditions obtained from the use of combined GA and spinal with NMB vs. the use of GA with spinal without NMB. 84 patients will all receive a single shot spinal and GA and then will be randomized to receive either NMB or placebo. The fracture reduction time will be measured.

DETAILED DESCRIPTION:
Eighty-four ASA I-IV patients presenting for operative repair of an unstable intertrochanteric femur fracture will be enrolled. This will include fractures classified according to the Orthopaedic Trauma Association / Arbeitsgemeinschaft fur Osteosynthesisfragen (OTA/AO) classification system as 31A2.2, 31A2.3, 31A3.1, 31A3.2, and 31A3.3.15 After consent and upon arrival to the operating room, patients will be monitored and then sedated with midazolam, fentanyl, and ketamine as necessary per standard practice to facilitate lateral positioning. Patients will be positioned with the operative side down for the spinal blockade. Under sterile conditions, spinal anesthesia will be induced with 10mg (1.2mL) of hyperbaric 0.75% bupivicaine as per standard practice. The patient will then be given a standard general anesthetic induction consisting of propofol, succinylcholine, fentanyl, and lidocaine. The patient will be intubated and anesthesia will be maintained with desflurane in oxygen and air. At the time of incision, the patient will be randomized to one of two groups. The surgeon and the anesthesiologist will be blinded to the patient's randomization status. Group 1 (NMB) will be given IV rocuronium 0.6mg/kg in a volume of 10cc. Group 2 (placebo) will be given 10cc normal saline. The anesthesia practitioner will test a Train of Four (TOF) and confirm a return of twitches prior to administering the study intervention. The nerve stimulator will then be disconnected until the conclusion of the case. Hemodynamic changes which suggest light anesthesia will be treated with additional fentanyl in 50mcg increments and/or increasing the desflurane concentration. Any hypotension directly attributed to the anesthetic by the anesthetic practitioner will be managed using a phenylephrine bolus and/or infusion as per standard anesthetic practice. Surgery will be performed by one of three fellowship trained orthopedic trauma surgeons, and fixation of these fractures will be with a single type of cephalomedullary implant (Synthes TFN-A, West Chester, PA). These three surgeons employ an identical bed, patient position, and traction technique (sterile skeletal traction) for these procedures. A percutaneous reduction will first be attempted. If unsuccessful, an open reduction will then be pursued. Following adequate reduction, fixation with the cephalomedullary implant will then be completed. Once skin closure has been initiated, to reverse any NMB, sugammadex 200mg in 2ml will be given to those patients randomized to the NMB group, and 2mL normal saline for the placebo group. At the discretion of the attending anesthesiologist, a nerve stimulator may be reapplied not less than 5 minutes after NMB reversal (or saline) is given. Once the attending surgeon has evaluated the final radiographs, all patients will have their anesthetics discontinued and will be extubated after emergence from anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-IV Age 55 or older Scheduled for operative repair of isolated intertrochanteric hip fracture

Exclusion Criteria:

* Inability to consent/refusal Allergy to any of the study medications Multiple traumatic injuries Contraindication to neuraxial or general anesthesia Pregnancy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Time to complete reduction of the fracture | Measured once Post-Op Day #0 in the recovery room
  Time necessary for complete reduction in the operating room.

SECONDARY OUTCOMES:
Surgical Operative Conditions | Measured once Post-Op Day #0 in the recovery room
  The surgeon's opinion of the operative conditions, as measured using a 4 point likert scale.
Estimated Blood Loss | Measured once Post-Op Day #0 in the recovery room
  Final estimated blood loss in mL for the procedure
Total operating room time | Measured once Post-Op Day #0 in the recovery room
  Total number of minutes spent in the operating room
Time to extubation | Measured once Post-Op Day #0 in the recovery room
  Total time from intubation to extubation
Intraoperative fentanyl use | Measured once Post-Op Day #0 in the recovery room
  Total amount (in mcg) of intravenous fentanyl used during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnell O, Kanis JA. An estimate of the worldwide prevalence and disability associated with osteoporotic fractures. Osteoporos Int. 2006 Dec;17(12):1726-33. doi: 10.1007/s00198-006-0172-4. Epub 2006 Sep 16. PMID 16983459
- [Background] Neuman MD, Silber JH, Elkassabany NM, Ludwig JM, Fleisher LA. Comparative effectiveness of regional versus general anesthesia for hip fracture surgery in adults. Anesthesiology. 2012 Jul;117(1):72-92. doi: 10.1097/ALN.0b013e3182545e7c. PMID 22713634
- [Background] Roche JJ, Wenn RT, Sahota O, Moran CG. Effect of comorbidities and postoperative complications on mortality after hip fracture in elderly people: prospective observational cohort study. BMJ. 2005 Dec 10;331(7529):1374. doi: 10.1136/bmj.38643.663843.55. Epub 2005 Nov 18. PMID 16299013
- [Background] Chu CC, Weng SF, Chen KT, Chien CC, Shieh JP, Chen JY, Wang JJ. Propensity Score-matched Comparison of Postoperative Adverse Outcomes between Geriatric Patients Given a General or a Neuraxial Anesthetic for Hip Surgery: A Population-based Study. Anesthesiology. 2015 Jul;123(1):136-47. doi: 10.1097/ALN.0000000000000695. PMID 25955981
- [Background] Basques BA, Bohl DD, Golinvaux NS, Samuel AM, Grauer JG. General versus spinal anaesthesia for patients aged 70 years and older with a fracture of the hip. Bone Joint J. 2015 May;97-B(5):689-95. doi: 10.1302/0301-620X.97B5.35042. PMID 25922465
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Bulka CM, Terekhov MA, Martin BJ, Dmochowski RR, Hayes RM, Ehrenfeld JM. Nondepolarizing Neuromuscular Blocking Agents, Reversal, and Risk of Postoperative Pneumonia. Anesthesiology. 2016 Oct;125(4):647-55. doi: 10.1097/ALN.0000000000001279. PMID 27496656
- [Background] Stewart PA, Liang SS, Li QS, Huang ML, Bilgin AB, Kim D, Phillips S. The Impact of Residual Neuromuscular Blockade, Oversedation, and Hypothermia on Adverse Respiratory Events in a Postanesthetic Care Unit: A Prospective Study of Prevalence, Predictors, and Outcomes. Anesth Analg. 2016 Oct;123(4):859-68. doi: 10.1213/ANE.0000000000001513. PMID 27537929
- [Background] Chang CC, Lin HC, Lin HW, Lin HC. Anesthetic management and surgical site infections in total hip or knee replacement: a population-based study. Anesthesiology. 2010 Aug;113(2):279-84. doi: 10.1097/ALN.0b013e3181e2c1c3. PMID 20657202
- [Background] Zorrilla-Vaca A, Grant MC, Mathur V, Li J, Wu CL. The Impact of Neuraxial Versus General Anesthesia on the Incidence of Postoperative Surgical Site Infections Following Knee or Hip Arthroplasty: A Meta-Analysis. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):555-63. doi: 10.1097/AAP.0000000000000437. PMID 27380106
- [Background] Mauermann WJ, Shilling AM, Zuo Z. A comparison of neuraxial block versus general anesthesia for elective total hip replacement: a meta-analysis. Anesth Analg. 2006 Oct;103(4):1018-25. doi: 10.1213/01.ane.0000237267.75543.59. PMID 17000823
- [Background] Minville V, Fourcade O, Grousset D, Chassery C, Nguyen L, Asehnoune K, Colombani A, Goulmamine L, Samii K. Spinal anesthesia using single injection small-dose bupivacaine versus continuous catheter injection techniques for surgical repair of hip fracture in elderly patients. Anesth Analg. 2006 May;102(5):1559-63. doi: 10.1213/01.ane.0000218421.18723.cf. PMID 16632842
- [Background] Mazze RI, Fujinaga M. Postdural puncture headache after continuous spinal anesthesia with 18-gauge and 20-gauge needles. Reg Anesth. 1993 Jan-Feb;18(1):47-51. PMID 8448099
- [Background] Holmstrom B, Laugaland K, Rawal N, Hallberg S. Combined spinal epidural block versus spinal and epidural block for orthopaedic surgery. Can J Anaesth. 1993 Jul;40(7):601-6. doi: 10.1007/BF03009695. PMID 8104724
- [Background] Marsh JL, Slongo TF, Agel J, Broderick JS, Creevey W, DeCoster TA, Prokuski L, Sirkin MS, Ziran B, Henley B, Audige L. Fracture and dislocation classification compendium - 2007: Orthopaedic Trauma Association classification, database and outcomes committee. J Orthop Trauma. 2007 Nov-Dec;21(10 Suppl):S1-133. doi: 10.1097/00005131-200711101-00001. PMID 18277234